CLINICAL TRIAL: NCT05248165
Title: Naples PCI Registry
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, MD, PhD, Federico II University
Other Study IDs: 232/18
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Myocardial Ischemia; Myocardial Infarction; Acute Coronary Syndrome
Keywords: Percutaneous coronary intervention; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary artery disease requiring percutaneous coronary intervention: Chronic or acute coronary syndrome requiring percutaneous myocardial revascularization.
  Interventions: Device: PCI

INTERVENTIONS:
Device: PCI — Percutaneous coronary intervention

SUMMARY:
The aim of the Naples PCI registry is to collect prospective data on baseline clinical, laboratory, and angiographic characteristics of patients undergoing PCI for acute or chronic coronary artery disease. All patients receive clinical follow-up at hospital discharge and at 1-year follow-up with the objective to assess clinical outcomes, including death, cardiovascular death, myocardial infarction, stroke, stent thrombosis, target-lesion and target-vessel revascularization, contrast-induced acute kidney injury, and bleeding events.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) constitutes the most commonly performed therapeutic procedure in cardiovascular medicine and one on the most frequent interventions performed in medicine. Since the introduction of the procedure more than 40 years ago, the safety and efficacy profile of PCI has steadily improved with continuous advances in the technique, equipment, and procedural success. In the late 1980s, the advent of coronary stents favored the widespread adoption of PCI in routine clinical practice by eliminating the risk of periprocedural abrupt closure related to coronary dissection and, as corollary, the need for standby emergent coronary artery bypass grafting. Nowadays, about three out of four patients requiring myocardial revascularization are managed PCI.

The objective of this study is to evaluate, within the framework of a prospective registry, the safety and efficacy of PCI by considering all device iterations including stent-based as well as non-stent-based interventions. We will evaluate clinical, laboratory, angiographic data of all patients undergoing PCI at the Federico II University Hospital. Clinical follow-up is collected during hospital stay and at 1-year after PCI. All adverse events are independently adjudicated by a clinical events committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical evidence of coronary artery disease requiring PCI;
2. Age ≥18 years;
3. Written informed consent.

Exclusion Criteria:

1. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease undergoing PCI at University of Naples "Federico II".
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2032-03-30 (Estimated); Study Completion 2032-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with death | 12 months
  Death
Number of patients with myocardial infarction | 12 months
  Myocardial infarction
Number of patients with stroke | 12 months
  Stroke
Number of patients with stent thrombosis | 12 months
  Stent thrombosis
Number of patients with target-vessel revascularization | 12 months
  Target vessel revascularization
Number of patients with target-lesion revascularization | 12 months
  Target lesion revascularization
Number of patients with contrast-induced acute kidney injury | 12 months
  Contrast-induced acute kidney injury
Number of patients with bleeding | 12 months
  Bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Advanced Biomedical Sciences, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piccolo R, Giustino G, Mehran R, Windecker S. Stable coronary artery disease: revascularisation and invasive strategies. Lancet. 2015 Aug 15;386(9994):702-13. doi: 10.1016/S0140-6736(15)61220-X. PMID 26334162
- [Background] Byrne RA, Stone GW, Ormiston J, Kastrati A. Coronary balloon angioplasty, stents, and scaffolds. Lancet. 2017 Aug 19;390(10096):781-792. doi: 10.1016/S0140-6736(17)31927-X. PMID 28831994
- [Background] Cuisset T, Verheugt FWA, Mauri L. Update on antithrombotic therapy after percutaneous coronary revascularisation. Lancet. 2017 Aug 19;390(10096):810-820. doi: 10.1016/S0140-6736(17)31936-0. PMID 28831996
- [Background] Rothwell PM. External validity of randomised controlled trials: "to whom do the results of this trial apply?". Lancet. 2005 Jan 1-7;365(9453):82-93. doi: 10.1016/S0140-6736(04)17670-8. PMID 15639683
- [Background] King M, Nazareth I, Lampe F, Bower P, Chandler M, Morou M, Sibbald B, Lai R. Impact of participant and physician intervention preferences on randomized trials: a systematic review. JAMA. 2005 Mar 2;293(9):1089-99. doi: 10.1001/jama.293.9.1089. PMID 15741531
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414